CLINICAL TRIAL: NCT01605734
Title: Phase II Trail of TACE Combinated With Sorafenib in Treating Patients With Unresectable Hepatocellular Carcinoma
Brief Title: TACE Combinated With Sorafenib in Treating Patients With Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinlong Song, Chief, Division of Interventiolal Therapy, Shandong Cancer Hospital and Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI-002
Record Dates: First submitted 2012-05-11; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: PHENYTOIN/SORAFENIB [VA Drug Interaction]; Carcinoma, Hepatocellular
Keywords: hepatocellular carcinoma; transarterial chemoembolization; sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group TACE (Active Comparator): TACE will be carried out with chemotherapeutic agents and lipiodol; additional embolisation will be carried out with gelatin sponge particles. TACE will be repeated if clinically indicated
  Interventions: Procedure: TACE
- Group Combination (Experimental): All patients will receive Sorafenib (800 mg/day) p.o. beginning four weeks after the first TACE and every day thereafter until patient death or premature withdrawal from study
  Interventions: Drug: sorafenib combined with TACE

INTERVENTIONS:
Procedure: TACE — After obtaining arterial access,a diagnostic visceral arteriogram will be performed to demonstrate arterial supply to the tumor and the presence of variant arterial anatomy.After having positioned the catheter within the artery feeding tumor,the chemoembolization mixture will be infused into th e artery until stagnant flow is observed.
  Arms: Group TACE
Drug: sorafenib combined with TACE — All patients will receive Sorafenib (800 mg/day) p.o. beginning four weeks after the first TACE and every day thereafter until patient death or premature withdrawal from study
  Arms: Group Combination

SUMMARY:
TACE is widely used in patients with unresectable HCC. However, it is a non-curative approach; thus ,strategies to further improve the survival of these patients are needed. Sorafenib is regarded as standard treatment for advanced HCC. It is the first systemic therapy to demonstrate a significant survival benefit in HCC patients.The hypothesis is that the combination of TACE with sorafenib could improve the survival of patients with unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed as HCC according to European Association for Study of the Liver criteria.
* BCLC stage B or C
* Child-Pugh class score≤8
* ECOG performance status ≤2
* Etiology: Hepatitis B virus(HBV) infection
* Written informed consent (approved by the Institutional Review Board [IRB]obtained prior to any study specific screening procedures
* Patient must be able to comply with the protocol
* Age 18-75 years
* Haematology:Absolute neutrophil count (ANC) > 1.5 x 109/L, Platelet count > 50 x 109/L, Haemoglobin > 9 g/dL (may be transfused to maintain or exceed this level) Prothrombin time international normalized ratio < 1.5
* Biochemistry:Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)< 5 x the upper limit of normal,Total bilirubin < 3 x the upper limit of normal,Serum creatinine < 1.5 x the upper limit of normal,Cholinesterase>0.5x the lower limit of normal，Prealbumin>0.5x the lower limit of normal.
* Life expectancy of > 3 months

Exclusion Criteria:

* BCLC stage D
* Child-Pugh Score≥9
* Clinically severe gastrointestinal bleeding within 4 weeks of the start of treatment
* Preexisting or history of hepatic encephalopathy
* uncontrolled hypertension
* Pregnancy (positive serum pregnancy test) or lactation
* Serious, non-healing wound, ulcer, or bone fracture
* Currently or recent (within the 30 days prior to starting study treatment) treatment of another investigational drug or participation in another investigational study
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents ( ≤ 6 months prior to study entry), myocardial infarction ( ≤ 6 months prior to study entry), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of Sorafenib/TACE or patient at high risk from treatment complications
* Other severe concomitant disease that may reduce life expectancy
* Risk of allergic reactions to the study drugs
* Drug abuse or other physical, psychological , or social problems that may interfere with the participation in the study or evaluation of study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Time to Progression | 1 year
  Time to progression is defined as time from randomization to radiological progression and will be evaluated every 8 week

SECONDARY OUTCOMES:
FACT-Hep | six months
  FACT-Hep is a chart established to evaluate the life quality of patients with HCC every 4 weeks
Disease control rate | six months after TACE
  CR+PR+SD
Safety | six months
  Number of participants with adverse events as a measure of safety and tolerability(According to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0)
PFS and OS | two years
  The overall survival is defined as time from randomization to death due to any cause, and will be evaluated every 8 weeks in the protocol treatment, and every one year in the follow-up period,respectively
Number of TACE sessions and the interval time between two TACE sessions | 2 years
AFP | six months

CONTACTS AND LOCATIONS:
Overall Officials: Jinlong Song, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (5):
- China (5):
  - Shandong Medical Imaging Research Institute, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - the Affiliated Hospital of Medical College Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong